CLINICAL TRIAL: NCT03401671
Title: A Phase 1, Open-label Study to Evaluate the Pharmacokinetics, Safety and Tolerability, and Pharmacodynamics of a Single Dose of Lanadelumab Administered Subcutaneously in Healthy Adult Japanese Subjects and Matched Healthy Adult Caucasian Subjects
Brief Title: Study of Lanadelumab in Healthy Japanese and Matched Caucasian Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHP643-101
Record Dates: First submitted 2018-01-10; First posted 2018-01-17 (Actual); Results first posted 2019-07-29 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers
Keywords: Lanadelumab
MeSH Terms: interventions — lanadelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Japanese (Experimental): Healthy subjects of Japanese descent will receive a single dose of 300 milligrams (mg) lanadelumab subcutaneous (SC) injection in the abdomen.
  Interventions: Drug: Lanadelumab
- Non-Hispanic Caucasians (Experimental): Healthy Non-Hispanic Caucasian subjects will receive a single dose of 300 mg lanadelumab SC injection in the abdomen
  Interventions: Drug: Lanadelumab

INTERVENTIONS:
Drug: Lanadelumab — SC injection of 300mg in 2mL (150 mg/mL) solution of lanadelumab will be administered as a single dose injection in the abdomen.
  Other Names: SHP643

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK), safety and tolerability and pharmacodynamics (PD) of lanadelumab in healthy adult Japanese subjects and matched non-Hispanic healthy adult Caucasian subjects.

ELIGIBILITY:
Inclusion Criteria:

* Ability to voluntarily provide written, signed, and dated informed consent as applicable to participate in the study.
* An understanding, ability, and willingness to fully comply with study procedures and restrictions.
* Age 18-55, inclusive, at the time of consent. The date of signature of the informed consent is defined as the beginning of the Screening Period. This inclusion criterion will only be assessed at the first screening visit.
* Subjects must be either:

  1. A subject of Japanese descent born in Japan, who has resided outside of Japan for no longer than 5 years and is of Japanese parentage, defined as having 2 Japanese parents and 4 Japanese grandparents, all born in Japan.
  2. A non-Hispanic, Caucasian subject who has 2 non-Hispanic, Caucasian parents and 4 non-Hispanic, Caucasian grandparents.
* Male or non-pregnant, non-lactating female who agrees to comply with any applicable contraceptive requirements of the protocol or females of non-childbearing potential.
* Considered "healthy" by the investigator. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, as well as a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, and urinalysis.
* Body mass index between 18.5-33 kilograms per square meter (kg/m^2), inclusive, with a body weight greater than or equal to (≥) 45 kg (99 pounds [lbs]). This inclusion criterion will only be assessed at the screening visit.
* Willing and able to consume standardized meals during the confinement period of the study. All subjects will be required to consume the identical meals on study days when serial PK and PD blood samples are collected.

Exclusion Criteria:

* History of any hematological, hepatic, respiratory, cardiovascular, renal, neurological or psychiatric disease, gall bladder removal, or current or recurrent disease that could affect the action, absorption, or disposition of the investigational product, or clinical or laboratory assessments.
* Current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to complete the study, or any condition that presents undue risk from the investigational product or procedures.
* Known or suspected intolerance or hypersensitivity to the investigational product, closely related compounds, or any of the stated ingredients.
* Significant illness, as judged by the investigator, within 2 weeks of the dose of investigational product.
* Known history of alcohol or other substance abuse within the last year, per the investigator.
* Donation of blood or blood products (example [e.g], plasma or platelets) within 60 days prior to receiving the dose of investigational product.
* Within 30 days prior to the dose of investigational product:

  1. Have used an investigational product (if elimination half-life is less than [<] 6 days, otherwise 5 half-lives).
  2. Have been enrolled in a clinical study (including vaccine studies) that, in the investigator's opinion, may impact this Shire-sponsored study.
* Confirmed systolic blood pressure (BP) greater than (>) 139 millimeter of mercury (mmHg) or <89mmHg, and diastolic BP >89mmHg or <49mmHg.
* Twelve-lead ECG values (average of triplicate readings) demonstrating QTc >450 milliseconds (msec) (males) or >470msec (females) at the Screening Visit or Day -1.
* Positive screen for drugs of abuse (that is, amphetamines, benzodiazepines, barbiturates, cocaine, marijuana, opiates, phencyclidine) at Screening, or drugs of abuse or alcohol on Day -1.
* Male subjects who consume more than 21 units of alcohol per week or 3 units per day. Female subjects who consume more than 14 units of alcohol per week or 2 units per day. One alcohol unit=1 beer or 1 wine (5 ounce [oz]/150 milliliter [mL]) or 1 liquor (1.5oz/40mL) or 0.75oz alcohol.
* Positive human immunodeficiency virus (HIV), hepatitis B virus surface antigen (HBsAg), or hepatitis C virus.(HCV) antibody screen.
* Use of tobacco in any form (eg, smoking or chewing) or other nicotine-containing products in any form (eg, gum, patch, electronic). Ex-users must report that they have stopped using tobacco for at least 30 days prior to receiving the dose of investigational product.
* Routine consumption of more than 2 units of caffeine per day or subjects who experience caffeine withdrawal headaches. One caffeine unit is contained in the following items: one 6oz (180mL) cup of coffee, two 12oz (360mL) cans of cola, one 12oz cup of tea, and three 1oz (85g) chocolate bars. Decaffeinated coffee, tea, or cola are not considered to contain caffeine.
* Current use of any medication (including over-the-counter, herbal, or homeopathic preparations; with the exception of hormonal replacement therapy or hormonal contraceptives). Current use is defined as use within 14 days of the dose of investigational product.
* Abnormal laboratory values considered clinically significant, as determined by the investigator at Screening or Day -1.
* History of any clinically significant surgery or procedure within 8 weeks of receiving the dose of investigational product, as determined by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- WCCT Global, Inc., Cypress, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in the United States between 15 January 2018 (first participant first visit) and 30 May 2018 (last participant last visit).
Pre-assignment Details: A total of 32 participants were enrolled, received the treatment and completed the study.
Groups:
- Japanese: Healthy participants of Japanese descent received a single dose of 300 milligrams (mg) lanadelumab subcutaneous (SC) injection in the abdomen.
- Non-Hispanic Caucasians: Healthy Non-Hispanic Caucasian participants received a single dose of 300 mg lanadelumab SC injection in the abdomen.
Period: Overall Study
Arm/Group | Japanese | Non-Hispanic Caucasians
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set consisted of all participants who received at least 1 dose of lanadelumab.
Groups:
- Japanese: Healthy participants of Japanese descent received a single dose of 300 mg lanadelumab SC injection in the abdomen.
- Total: Total of all reporting groups
Arm/Group | Japanese | Non-Hispanic Caucasians | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.4 (7.82) | 42.8 (6.40) | 43.1 (7.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 16 | 0 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 16 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Lanadelumab
Description: Cmax is the maximum observed plasma concentration of Lanadelumab was presented. Geometric mean and geometric coefficient of variation percent (CV%) was presented.
Time Frame: Pre-dose, 8, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344, 2016 and 2688 hours post-dose
Population: Pharmacokinetic (PK) set consisted of all participants who received at least 1 dose of lanadelumab and had at least 1 evaluable post-dose PK concentration value.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (ug/mL)
Arm/Group | Japanese | Non-Hispanic Caucasians
Number analyzed (Participants) | 16 | 16
microgram per milliliter (ug/mL) | 21.91 (38) | 21.42 (25)
Statistical Analysis 1: Comparison: Japanese vs Non-Hispanic Caucasians; An analysis of variance was performed with the natural log-transformed PK parameters as the dependent variable and ethnic group as a fixed effect; Test type: Other — Analysis was performed for estimation of least square means only. Descriptive statistical analysis was the main analysis; Ratio of Geometric least squares Means = 1.0229, 90% CI 2-sided [0.8473 to 1.2349]

2. Primary Outcome: Time to Reach Maximum Observed Drug Concentration in Plasma (Tmax) of Lanadelumab
Description: Tmax of Lanadelumab was presented.
Time Frame: Pre-dose, 8, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344, 2016 and 2688 hours post-dose
Population: PK set consisted of all participants who received at least 1 dose of lanadelumab and had at least 1 evaluable post-dose PK concentration value.
Measure: Median (Full Range); unit: day
Arm/Group | Japanese | Non-Hispanic Caucasians
Number analyzed (Participants) | 16 | 16
day | 5.67 [2.00 to 6.11] | 5.00 [3.00 to 13.00]

3. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUC0-last) in Plasma of Lanadelumab
Description: AUC(0-last) of Lanadelumab was presented. Geometric mean and geometric coefficient of variation percent (CV%) was presented.
Time Frame: Pre-dose, 8, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344, 2016 and 2688 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*microgram per milliliter(day*ug/mL)
Arm/Group | Japanese | Non-Hispanic Caucasians
Number analyzed (Participants) | 16 | 16
day*microgram per milliliter(day*ug/mL) | 510.6 (30) | 547.6 (20)
Statistical Analysis 1: Comparison: Japanese vs Non-Hispanic Caucasians; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of Geometric least squares Means = 0.9324, 90% CI 2-sided [0.8016 to 1.0846]

4. Primary Outcome: Area Under the Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Lanadelumab
Description: AUC(0-infinity) of Lanadelumab was presented.Geometric mean and geometric coefficient of variation percent (CV%) was presented.
Time Frame: Pre-dose, 8, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344, 2016 and 2688 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*microgram per milliliter(day* ug/mL)
Arm/Group | Japanese | Non-Hispanic Caucasians
Number analyzed (Participants) | 16 | 16
day*microgram per milliliter(day* ug/mL) | 515.0 (30) | 552.7 (20)
Statistical Analysis 1: Comparison: Japanese vs Non-Hispanic Caucasians; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of Geometric least squares Means = 0.9318, 90% CI 2-sided [0.8005 to 1.0846]

5. Primary Outcome: Terminal Elimination Rate Constant (Lambda z) for Lanadelumab
Description: Lambda z of Lanadelumab was presented.Geometric mean and geometric coefficient of variation percent (CV%) was presented.
Time Frame: Pre-dose, 8, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344, 2016 and 2688 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: per day
Arm/Group | Japanese | Non-Hispanic Caucasians
Number analyzed (Participants) | 16 | 16
per day | 0.04470 (9) | 0.04385 (11)

6. Primary Outcome: Terminal Half-life (t12) of Lanadelumab
Description: t1/2 of Lanadelumab was presented.
Time Frame: Pre-dose, 8, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344, 2016 and 2688 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: day
Arm/Group | Japanese | Non-Hispanic Caucasians
Number analyzed (Participants) | 16 | 16
day | 15.54 [12.8 to 17.9] | 15.59 [12.4 to 19.1]

7. Primary Outcome: Apparent Clearance (CL/F) of Lanadelumab
Description: CL/F of Lanadelumab was presented.Geometric mean and geometric coefficient of variation percent (CV%) was presented.
Time Frame: Pre-dose, 8, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344, 2016 and 2688 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per day
Arm/Group | Japanese | Non-Hispanic Caucasians
Number analyzed (Participants) | 16 | 16
liter per day | 0.5826 (30) | 0.5428 (20)

8. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Lanadelumab
Description: Vz/F of Lanadelumab was presented.Geometric mean and geometric coefficient of variation percent (CV%) was presented.
Time Frame: Pre-dose, 8, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344, 2016 and 2688 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Japanese | Non-Hispanic Caucasians
Number analyzed (Participants) | 16 | 16
liter | 13.03 (29) | 12.38 (22)

9. Primary Outcome: Body-weight Adjusted Area Under the Concentration-Time Curve From Time Zero to the Last Quantifiable Concentration (AUC0-last) in Plasma of Lanadelumab
Description: Body-weight adjusted AUC(0-last) of Lanadelumab was presented. Geometric mean and geometric coefficient of variation percent (CV%) was presented.
Time Frame: Pre-dose, 8, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344, 2016 and 2688 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL/kg
Arm/Group | Japanese | Non-Hispanic Caucasians
Number analyzed (Participants) | 16 | 16
day*ug/mL/kg | 510.6 (30) | 547.6 (20)

10. Primary Outcome: Body-weight Adjusted Area Under the Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) in Plasma of Lanadelumab
Description: Body-weight adjusted AUC(0-infinity) of Lanadelumab was presented. Geometric mean and geometric coefficient of variation percent (CV%) was presented.
Time Frame: Pre-dose, 8, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344, 2016 and 2688 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL/kg
Arm/Group | Japanese | Non-Hispanic Caucasians
Number analyzed (Participants) | 16 | 16
day*ug/mL/kg | 8.012 (44) | 7.950 (27)

11. Primary Outcome: Body-weight Adjusted Maximum Observed Plasma Concentration (Cmax) of Lanadelumab
Description: Body-weight adjusted Cmax of Lanadelumab was presented.Geometric mean and geometric coefficient of variation percent (CV%) was presented.
Time Frame: Pre-dose, 8, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344, 2016 and 2688 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: microgram per milliliter per kilogram
Arm/Group | Japanese | Non-Hispanic Caucasians
Number analyzed (Participants) | 16 | 16
microgram per milliliter per kilogram | 0.3236 [0.125 to 0.722] | 0.3042 [0.196 to 0.709]

12. Primary Outcome: Body-weight Adjusted Apparent Clearance (CL/F) of Lanadelumab
Description: Body-weight adjusted CL/F of Lanadelumab was presented.Geometric mean and geometric coefficient of variation percent (CV%) was presented.
Time Frame: Pre-dose, 8, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344, 2016 and 2688 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per day per kilogram (L/day/kg)
Arm/Group | Japanese | Non-Hispanic Caucasians
Number analyzed (Participants) | 16 | 16
liter per day per kilogram (L/day/kg) | 0.009064 (23) | 0.007809 (20)

13. Primary Outcome: Body-weight Adjusted Apparent Volume of Distribution (Vz/F) of Lanadelumab
Description: Body-weight adjusted Vz/F of Lanadelumab was presented.Geometric mean and geometric coefficient of variation percent (CV%) was presented.
Time Frame: Pre-dose, 8, 24, 48, 72, 96, 168, 336, 504, 672, 1008, 1344, 2016 and 2688 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per kilogram (L/kg)
Arm/Group | Japanese | Non-Hispanic Caucasians
Number analyzed (Participants) | 16 | 16
liter per kilogram (L/kg) | 0.2028 (23) | 0.1781 (20)

14. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Based on Severity, Seriousness and Causality
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation participants administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. TEAEs are defined as AEs with onset at the time of or following the first exposure to study drug, or medical conditions present prior to the start of study drug but increasing in severity or relationship at the time of or following the start of treatment, up to the last follow-up visit. Severity of an AE is determined by following definitions: Mild: An event that does not generally interfere with usual activities of daily living; Moderate: An event that interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the research participants; Severe: An AE that interrupts usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention.
Time Frame: From start of study drug administration up to follow-up (up to 115 days)
Population: Safety analysis set included all participants who received at least 1 dose of Lanadelumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Japanese | Non-Hispanic Caucasians
Number analyzed (Participants) | 16 | 16
Participants
  Participants with Mild TEAE | 6 | 4
  Participants with Moderate TEAE | 1 | 5
  Participants with Severe TEAE | 0 | 0
  Participants with Serious TEAE | 0 | 0
  Participants with Non-Serious TEAE | 7 | 9
  Participants with Causality (Death) | 0 | 0

15. Secondary Outcome: Number of Participants With Clinically Significant Change in Clinical Laboratory Results Reported as an Adverse Event
Description: Clinical laboratory assessments include hematology, clinical chemistry, coagulation and urinalysis. The investigator will assess out-of-range clinical laboratory values for clinical significance, to indicate whether or not the values are clinically significant. Any changes from baseline in clinical laboratory results which are deemed clinically significant by the investigator are to be recorded as an AE.
Time Frame: From start of study drug administration up to follow-up (up to 115 days)
Population: Safety analysis set included all participants who received at least 1 dose of Lanadelumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Japanese | Non-Hispanic Caucasians
Number analyzed (Participants) | 16 | 16
Participants | 0 | 0

16. Secondary Outcome: Number of Participants With Clinically Significant Change in Vital Signs Reported as an Adverse Event
Description: Vital sign assessments include blood pressure, pulse rate and body temperature. Any changes from baseline in vital signs which are deemed clinically significant by the investigator are to be recorded as an AE.
Time Frame: From start of study drug administration up to follow-up (up to 115 days)
Population: Safety analysis set included all participants who received at least 1 dose of Lanadelumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Japanese | Non-Hispanic Caucasians
Number analyzed (Participants) | 16 | 16
Participants | 0 | 0

17. Secondary Outcome: Number of Participants With Clinically Significant Change in Electrocardiogram (ECG) Reported as an Adverse Event
Description: Twelve-lead ECG will be performed after 5 minutes of rest in the supine position. Any change in ECG assessments which are deemed clinically significant by the investigator are to be reported as AE.
Time Frame: From start of study drug administration up to follow-up (up to 115 days)
Population: Safety analysis set includes all participants who received at least 1 dose of Lanadelumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Japanese | Non-Hispanic Caucasians
Number analyzed (Participants) | 16 | 16
Participants | 0 | 0

18. Secondary Outcome: Number of Participants Who Developed Antidrug Antibodies to Lanadelumab at Specified Time Points
Description: Plasma samples were analyzed for presence of antidrug antibodies to lanadelumab. Participants who show positive results for lanadelumab antibodies were reported.
Time Frame: Day 1, 14, 28, 56, and 112 (End of Study/Early Termination [EOS/ET])
Population: Safety analysis set included all participants who received at least 1 dose of lanadelumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Japanese | Non-Hispanic Caucasians
Number analyzed (Participants) | 16 | 16
Participants
  Participants with positive ADA: Day 1 | 0 | 0
  Participants with positive ADA: Day 14 | 0 | 0
  Participants with positive ADA: Day 28 | 0 | 0
  Participants with positive ADA: Day 56 | 0 | 0
  Participants with positive ADA: Day 112 (EOS/ET) | 0 | 1

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow-up (up to 115 days)
Arm/Group | Japanese | Non-Hispanic Caucasians
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 7/16 | 9/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Japanese (N=16) | Non-Hispanic Caucasians (N=16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Injection site erythema (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (3)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT03401671/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/71/NCT03401671/SAP_001.pdf